CLINICAL TRIAL: NCT01415427
Title: A Multicenter, Multinational, Extension Study to Evaluate the Long-Term Efficacy and Safety of BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Brief Title: Long-Term Efficacy and Safety Extension Study of BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR-005
Record Dates: First submitted 2011-08-08; First posted 2011-08-12 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2017-04

CONDITIONS: Mucopolysaccharidosis IV A; Morquio A Syndrome; MPS IVA
Keywords: Mucopolysaccharidosis IV type A; MPS IV Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — Chondroitinases and Chondroitin Lyases; Galns protein, mouse; GALNS protein, human; Enzyme Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMN 110 Weekly (Experimental): BMN 110 Weekly: In Part 1, patients will receive an intravenous infusion of BMN 110 at a dose of 2.0 mg/kg administered over a period of approximately 4 hours once a week.
  Interventions: Drug: BMN 110 - Weekly
- BMN 110 Every Other Week (Experimental): BMN 110 Every Other Week: In Part 1, patients will receive an intravenous infusion of BMN 110 at a dose of 2.0 mg/kg administered over a period of approximately 4 hours every other week and will receive infusions of placebo on alternating weeks.
  Interventions: Drug: BMN 110 - Every Other Week

INTERVENTIONS:
Drug: BMN 110 - Weekly — In Part 1, patients will receive intravenous (IV) infusions of study drug at a dose of 2.0 mg/kg/qw administered over a period of approximately 4 hours once a week.
  In Part 2, patients will continue to receive 2.0 mg/kg of BMN 110 every week, with no placebo.
  Other Names: N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
  Arms: BMN 110 Weekly
Drug: BMN 110 - Every Other Week — In Part 1, patients will receive intravenous (IV) infusions of study drug at a dose of 2.0 mg/kg administered over a period of approximately 4 hours every other week. Patients randomized to the 2.0 mg/kg/qow arm will receive infusions of placebo on alternating weeks, to mask active drug weeks.
  In Part 2, patients will receive 2.0 mg/kg of BMN 110 every week, with no placebo.
  Other Names: N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
  Arms: BMN 110 Every Other Week

SUMMARY:
This Phase 3 extension study will evaluate the long-term efficacy and safety of BMN 110 2.0 mg/kg/week and/or BMN 110 2.0 mg/kg/every other week in patients with mucopolysaccharidosis IVA (Morquio A Syndrome).

DETAILED DESCRIPTION:
This is a multi-center, multinational, extension study to evaluate 2 dose regimens of BMN 110 treatment in patients with MPS IVA who completed MOR-004.

The last study visit assessments for MOR-004 will constitute Baseline for this study. The first study drug dose of this protocol will occur on Week 0 of MOR-005, which is the same as the last visit (Week 24) of MOR-004. Initially, the study will be double-blind with patients previously randomized to BMN 110 in MOR-004 remaining on their assigned BMN 110 dose regimen (qw or qow dosing). The MOR-004 placebo patients will be re-randomized (1:1 ratio) to one of the 2 BMN 110 dose regimen groups: 2.0 mg/kg/qw or 2.0 mg/kg/qow.

There will be two study parts:

* Part 1 - randomized double-blind until the optimal BMN 110 dose regimen has been determined, based on the final primary efficacy analysis from MOR-004
* Part 2 - open-label BMN 110 treatment with the single optimal dose regimen

ELIGIBILITY:
Inclusion Criteria:

* Must have completed MOR-004
* Is willing and able to provide written, signed informed consent. Or in the case of patients under the age of 18 (or other age as defined by regional law or regulation), provide written assent (if required) and have written informed consent, signed by a legally authorize representative, after the nature of the study has been explained, and prior to performance of research-related procedures.
* If sexually active, must be willing to use an acceptable method of contraception while participating in the study.
* If female, of childbearing potential, must have a negative pregnancy test at Baseline and be willing to have additional pregnancy tests done during the study.

Exclusion Criteria:

* Is pregnant or breastfeeding, at Baseline, or planning to become pregnant (self or partner) at any time during the study.
* Has used any investigational product (other than BMN 110 in MOR-004), or investigational medical device, within 30 days prior to Baseline; or is required to use any investigational agent prior to completion of all scheduled study assessments.
* Was enrolled in a previous BMN 110 study, other than MOR-004.
* Has a concurrent disease or condition, including but not limited to, symptomatic cervical spine instability, clinically significant spinal cord compression, or severe cardiac disease that would interfere with study participation, or pose a safety risk, as determined by the Investigator.
* Has any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2011-07; Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lounsbury, Study Director — BioMarin Pharmaceutical
Locations (39):
- United States (10):
  - Phoenix, Arizona
  - Oakland, California
  - Orange, California
  - Wilmington, Delaware
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - New York, New York
  - Seattle, Washington
- Córdoba, Argentina
- Brazil (3):
  - Campina Grande
  - Porto Alegre
  - Rio de Janeiro
- Canada (3):
  - Montreal
  - Sherbrooke
  - Toronto
- Bogotá, Colombia
- Copenhagen, Denmark
- France (3):
  - Lyon
  - Marseille
  - Paris
- Mainz, Germany
- Monza, Italy
- Tokyo, Japan
- Amsterdam, Netherlands
- Oslo, Norway
- Portugal (2):
  - Coimbra
  - Lisbon
- Doha, Qatar
- Riyadh, Saudi Arabia
- Seoul, South Korea
- Santiago de Compostela, Spain
- Taipei, Taiwan
- Ankara, Turkey (Türkiye)
- United Kingdom (4):
  - Belfast
  - Birmingham
  - London
  - Manchester

REFERENCES:
- [Derived] Hendriksz CJ, Parini R, AlSayed MD, Raiman J, Giugliani R, Mitchell JJ, Burton BK, Guelbert N, Stewart FJ, Hughes DA, Matousek R, Hawley SM, Decker C, Harmatz PR. Impact of long-term elosulfase alfa on activities of daily living in patients with Morquio A syndrome in an open-label, multi-center, phase 3 extension study. Mol Genet Metab. 2018 Feb;123(2):127-134. doi: 10.1016/j.ymgme.2017.11.015. Epub 2017 Dec 5. PMID 29248359
- [Derived] Hughes D, Giugliani R, Guffon N, Jones SA, Mengel KE, Parini R, Matousek R, Hawley SM, Quartel A. Clinical outcomes in a subpopulation of adults with Morquio A syndrome: results from a long-term extension study of elosulfase alfa. Orphanet J Rare Dis. 2017 May 23;12(1):98. doi: 10.1186/s13023-017-0634-0. PMID 28535791
- [Derived] Long B, Tompkins T, Decker C, Jesaitis L, Khan S, Slasor P, Harmatz P, O'Neill CA, Schweighardt B. Long-term Immunogenicity of Elosulfase Alfa in the Treatment of Morquio A Syndrome: Results From MOR-005, a Phase III Extension Study. Clin Ther. 2017 Jan;39(1):118-129.e3. doi: 10.1016/j.clinthera.2016.11.017. Epub 2016 Dec 10. PMID 27955919

RESULTS

PARTICIPANT FLOW:
Groups:
- PBO-QOW: Weekly IV infusions of placebo solution for a total of 24 consecutive weeks in MOR004 + Biweekly infusions of 2.0 mg/kg/qow BMN 110 and infusions of placebo on alternating weeks in MOR005
- PBO-QW: Weekly IV infusions of placebo solution for a total of 24 consecutive weeks in MOR004 +Weekly infusions of 2.0 mg/kg/week BMN 110 in MOR005
- QOW-QOW: Biweekly infusions of 2.0 mg/kg/qow BMN 110 and infusions of placebo on alternating weeks for a total of 24 consecutive weeks in MOR004 + Biweekly infusions of 2.0 mg/kg/qow BMN 110 and infusions of placebo on alternating weeks in MOR005
- QW-QW: Weekly infusions of 2.0 mg/kg/week BMN 110 for a total of 24 consecutive weeks in MOR004 + Weekly infusions of 2.0 mg/kg/week BMN 110 in MOR005
Period: Overall Study
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW
Started | 29 | 29 | 59 | 56
Completed | 0 | 0 | 1 | 0
Not Completed | 29 | 29 | 58 | 56

BASELINE CHARACTERISTICS:
Groups:
- PBO-QOW: Placebo in MOR004 + BMN110 2.0 mg/kg/qow in MOR005
- PBO-QW: Placebo in MOR004 + BMN110 2.0 mg/kg/qw in MOR005
- QOW-QOW: BMN110 2.0 mg/kg/qow in MOR004 + BMN110 2.0 mg/kg/qow in MOR005
- QW-QW: BMN110 2.0 mg/kg/qw in MOR004 + BMN110 2.0 mg/kg/qw in MOR005
- Total: Total of all reporting groups
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
Number analyzed (Participants) | 29 | 29 | 59 | 56 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (13.66) | 13.5 (8.50) | 15.3 (10.79) | 12.8 (8.01) | 14.4 (10.20)
Age, Customized [Number; unit: participants]
  5 - 11 | 15 | 15 | 31 | 32 | 93
  12 - 18 | 7 | 7 | 16 | 16 | 46
  >=19 | 7 | 7 | 12 | 8 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 25 | 30 | 87
  Male | 15 | 11 | 34 | 26 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 16 | 9 | 37
  Not Hispanic or Latino | 25 | 21 | 43 | 47 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 7 | 15 | 14 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2 | 4
  White | 25 | 18 | 35 | 35 | 113
  Other | 0 | 4 | 7 | 5 | 16
Region of Enrollment [Number; unit: participants]
  Argentina | 0 | 1 | 1 | 0 | 2
  Brazil | 2 | 3 | 10 | 5 | 20
  Canada | 3 | 1 | 5 | 5 | 14
  Colombia | 0 | 2 | 2 | 2 | 6
  Denmark | 0 | 0 | 0 | 1 | 1
  France | 2 | 5 | 5 | 8 | 20
  Germany | 2 | 2 | 5 | 1 | 10
  Italy | 3 | 1 | 4 | 2 | 10
  Japan | 0 | 0 | 4 | 2 | 6
  Korea, South | 2 | 1 | 1 | 3 | 7
  Netherlands | 1 | 0 | 2 | 3 | 6
  Portugal | 1 | 1 | 1 | 0 | 3
  Qatar | 0 | 1 | 0 | 1 | 2
  Saudi Arabia | 0 | 2 | 1 | 4 | 7
  Taiwan | 0 | 1 | 3 | 1 | 5
  United Kingdom | 6 | 3 | 4 | 9 | 22
  United States | 7 | 5 | 11 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6-minute Walk (6MW) Test - ITT
Description: Efficacy was assessed by changes from baseline in 6-minute walk test
Time Frame: Baseline to week 168
Population: ITT-intent-to-treat population, defined as all patients enrolled in the study who received patient IDs regardless of whether they received study drug or not.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Total: All treatment groups
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
Number analyzed (Participants) | 29 | 29 | 59 | 58 | 176
meters
  Baseline | 219.7 (74.22) | 207.2 (64.87) | 205.7 (81.19) | 203.9 (76.32) | 207.2 (75.58)
  Change from Baseline to Week 24: number analyzed (Participants) | 29 | 29 | 59 | 57 | 175
  Change from Baseline to Week 24 | 23.8 (56.21) | 5.0 (43.27) | 11.1 (49.95) | 36.5 (58.49) | 20.2 (54.02)
  Change from Baseline to Week 72: number analyzed (Participants) | 28 | 27 | 57 | 55 | 167
  Change from Baseline to Week 72 | 41.5 (89.24) | -1.5 (112.07) | 27.2 (56.66) | 30.6 (73.66) | 26.1 (79.26)
  Change from Baseline to Week 120: number analyzed (Participants) | 28 | 27 | 54 | 54 | 163
  Change from Baseline to Week 120 | 32.3 (92.13) | -2.9 (95.69) | 6.0 (86.28) | 29.7 (81.37) | 16.9 (87.67)
  Change from Baseline to Week 168: number analyzed (Participants) | 10 | 13 | 32 | 26 | 81
  Change from Baseline to Week 168 | 52.2 (100.07) | 20.1 (80.79) | 5.2 (81.54) | -8.8 (101.24) | 8.9 (90.81)

2. Primary Outcome: Change From Baseline in 6-minute Walk (6MW) Test - MPP
Description: Efficacy was assessed by changes from baseline in 6-minute walk test
Time Frame: Baseline to week 168
Population: MPP- modified per-protocol population, define as the ITT(intent to treat) after removing patients who had orthosurgery in first 120 weeks or <96 doses in first 120 weeks.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
Number analyzed (Participants) | 20 | 19 | 42 | 43 | 124
meters
  Baseline | 208.7 (78.12) | 190.2 (65.54) | 195.9 (80.40) | 208.8 (73.24) | 201.6 (74.94)
  Change from Baseline to Week 24 | 30.3 (56.53) | 9.6 (46.87) | 13.6 (52.65) | 41.5 (59.89) | 25.4 (56.08)
  Change from Baseline to Week 72: number analyzed (Participants) | 20 | 18 | 42 | 43 | 123
  Change from Baseline to Week 72 | 54.5 (85.19) | 37.7 (69.35) | 35.3 (58.19) | 37.5 (72.17) | 39.6 (69.11)
  Change from Baseline to Week 120: number analyzed (Participants) | 20 | 19 | 41 | 43 | 123
  Change from Baseline to Week 120 | 60.8 (64.45) | 19.8 (86.69) | 19.7 (77.29) | 38.6 (66.65) | 33.0 (73.94)
  Change from Baseline to Week 168: number analyzed (Participants) | 5 | 8 | 26 | 22 | 61
  Change from Baseline to Week 168 | 85.8 (128.04) | 14.6 (94.41) | 10.0 (84.66) | -12.3 (106.34) | 8.8 (98.69)

3. Secondary Outcome: Change From Baseline in 3-minute Stair Climb Test - ITT
Description: Efficacy was assessed by changes from baseline in 3-minute stair climb test.
Time Frame: Baseline to week 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: stairs/min
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
Number analyzed (Participants) | 29 | 29 | 59 | 58 | 176
stairs/min
  Baseline | 33.1 (15.60) | 26.9 (12.08) | 27.1 (15.80) | 29.6 (16.44) | 28.9 (15.42)
  Change from Baseline to Week 24: number analyzed (Participants) | 29 | 29 | 59 | 57 | 175
  Change from Baseline to Week 24 | 4.7 (9.65) | 2.9 (7.30) | 2.9 (10.94) | 4.8 (8.06) | 3.8 (9.25)
  Change from Baseline to Week 72: number analyzed (Participants) | 28 | 26 | 56 | 54 | 164
  Change from Baseline to Week 72 | 8.9 (15.44) | 1.2 (14.95) | 5.5 (11.96) | 5.3 (9.88) | 5.3 (12.60)
  Change from Baseline to Week 120: number analyzed (Participants) | 28 | 27 | 54 | 53 | 162
  Change from Baseline to Week 120 | 6.0 (17.05) | 1.7 (14.80) | 4.7 (14.60) | 5.8 (13.42) | 4.8 (14.65)
  Change from baseline to week 168: number analyzed (Participants) | 10 | 13 | 32 | 25 | 80
  Change from baseline to week 168 | 8.9 (17.57) | 5.5 (15.44) | 4.6 (13.64) | 0.4 (20.96) | 4.0 (16.90)

4. Secondary Outcome: Change From Baseline in 3-minute Stair Climb Test - MPP
Description: Efficacy was assessed by changes from baseline in 3-minute stair climb test.
Time Frame: Baseline to week 168
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: stairs/min
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
Number analyzed (Participants) | 20 | 19 | 42 | 43 | 124
stairs/min
  Baseline | 33.1 (14.12) | 24.8 (13.92) | 25.6 (13.73) | 31.3 (16.22) | 28.7 (14.93)
  Change from Baseline to Week 24 | 3.4 (8.09) | 3.6 (8.63) | 5.0 (11.46) | 3.9 (7.67) | 4.1 (9.23)
  Change from Baseline to Week 72: number analyzed (Participants) | 20 | 18 | 42 | 43 | 123
  Change from Baseline to Week 72 | 10.4 (13.77) | 6.1 (10.56) | 7.4 (12.53) | 5.7 (9.98) | 7.1 (11.61)
  Change from Baseline to Week 120: number analyzed (Participants) | 20 | 19 | 41 | 42 | 122
  Change from Baseline to Week 120 | 9.1 (13.38) | 4.2 (12.49) | 8.1 (13.83) | 7.2 (12.58) | 7.4 (13.05)
  Change from baseline to week 168: number analyzed (Participants) | 5 | 8 | 26 | 21 | 60
  Change from baseline to week 168 | 12.4 (23.03) | 4.3 (17.82) | 6.0 (14.59) | -2.6 (18.47) | 3.3 (17.39)

5. Secondary Outcome: Change From Baseline in Urine Keratan Sulfate - ITT
Description: Efficacy was assessed by changes from baseline in urine keratan sulfate (normalized to urine creatinine.)
Time Frame: Baseline to week 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mg
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
Number analyzed (Participants) | 29 | 29 | 59 | 58 | 176
ug/mg
  Baseline: number analyzed (Participants) | 28 | 29 | 59 | 58 | 176
  Baseline | 22.7 (15.27) | 28.5 (14.89) | 28.6 (21.17) | 26.9 (14.11) | 27.1 (17.05)
  Percent Change from Baseline to Week 24: number analyzed (Participants) | 26 | 28 | 57 | 54 | 166
  Percent Change from Baseline to Week 24 | 3.4 (29.15) | -11.3 (23.68) | -35.2 (20.70) | -45.1 (19.89) | -28.2 (28.46)
  Percent Change from Baseline to Week 72: number analyzed (Participants) | 26 | 28 | 57 | 51 | 162
  Percent Change from Baseline to Week 72 | -54.1 (17.21) | -56.8 (13.69) | -55.6 (14.23) | -53.7 (17.45) | -55.0 (15.61)
  Percent Change from Baseline to Week 120: number analyzed (Participants) | 26 | 24 | 53 | 53 | 156
  Percent Change from Baseline to Week 120 | -55.5 (18.60) | -62.2 (15.39) | -55.8 (26.56) | -61.5 (20.59) | -58.7 (21.88)
  Percent Change from Baseline to Week 168: number analyzed (Participants) | 8 | 11 | 27 | 18 | 64
  Percent Change from Baseline to Week 168 | -31.9 (31.20) | -38.3 (47.43) | -28.5 (35.14) | -39.3 (47.39) | -33.7 (40.06)

6. Secondary Outcome: Change From Baseline in Urine Keratan Sulfate - MPP
Description: Efficacy was assessed by changes from baseline in urine keratan sulfate (normalized to urine creatinine.)
Time Frame: Baseline to week 168
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/mg
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
Number analyzed (Participants) | 20 | 19 | 42 | 43 | 124
ug/mg
  Baseline: number analyzed (Participants) | 19 | 19 | 42 | 43 | 123
  Baseline | 21.2 (15.55) | 27.5 (15.24) | 27.2 (22.90) | 24.9 (13.13) | 25.5 (17.61)
  Percent Change from Baseline to Week 24: number analyzed (Participants) | 17 | 19 | 41 | 40 | 117
  Percent Change from Baseline to Week 24 | 1.2 (24.34) | -12.9 (24.29) | -35.5 (22.62) | -44.9 (19.60) | -29.7 (27.52)
  Percent Change from Baseline to Week 72: number analyzed (Participants) | 18 | 19 | 41 | 41 | 119
  Percent Change from Baseline to Week 72 | -51.7 (19.34) | -58.8 (14.60) | -56.9 (13.55) | -53.7 (17.87) | -55.3 (16.21)
  Percent Change from Baseline to Week 120: number analyzed (Participants) | 18 | 17 | 40 | 42 | 117
  Percent Change from Baseline to Week 120 | -58.3 (15.87) | -64.2 (16.58) | -62.1 (15.97) | -61.8 (21.28) | -61.7 (17.98)
  Percent Change from Baseline to Week 168: number analyzed (Participants) | 4 | 7 | 22 | 15 | 48
  Percent Change from Baseline to Week 168 | -9.9 (23.48) | -41.6 (46.05) | -27.1 (37.28) | -43.0 (34.07) | -32.8 (37.11)

ADVERSE EVENTS:
Time Frame: Study Period
Groups:
- PBO-QOW: PBO-QOW
- PBO-QW: PBO-QW
- QOW-QOW: QOW-QOW
- QW-QW: QW-QW
- Total: Total
Arm/Group | PBO-QOW | PBO-QW | QOW-QOW | QW-QW | Total
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 1/59 | 0/56 | 1/173
Serious Adverse Events (participants affected / at risk) | 17/29 | 15/29 | 26/59 | 31/56 | 89/173
Other Adverse Events (participants affected / at risk) | 29/29 | 29/29 | 59/59 | 56/56 | 173/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBO-QOW (N=29) | PBO-QW (N=29) | QOW-QOW (N=59) | QW-QW (N=56) | Total (N=173)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Congenital osteodystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 4 (6)
Device dislocation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Mononucleosis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (4)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Joint instability (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Knee deformity (Musculoskeletal and connective tissue disorders) | 6 (8) | 8 (9) | 7 (7) | 8 (8) | 29 (32)
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Spinal cord ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somatoform disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Child abuse (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 5 (5)
Epiphyseal stapling (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Poor venous access (Vascular disorders) | 0 (0) | 2 (2) | 5 (5) | 5 (5) | 12 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBO-QOW (N=29) | PBO-QW (N=29) | QOW-QOW (N=59) | QW-QW (N=56) | Total (N=173)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Aortic valve disease (Cardiac disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 9 (9)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 3 (3) | 8 (8) | 4 (4) | 16 (16)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Mitral valve disease (Cardiac disorders) | 1 (1) | 1 (1) | 6 (6) | 3 (4) | 11 (12)
Mitral valve incompetence (Cardiac disorders) | 4 (4) | 6 (6) | 12 (12) | 4 (5) | 26 (27)
Palpitations (Cardiac disorders) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 6 (8)
Pulmonary valve incompetence (Cardiac disorders) | 2 (2) | 3 (3) | 2 (2) | 5 (5) | 12 (12)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (11) | 6 (17)
Tachycardia (Cardiac disorders) | 8 (14) | 4 (15) | 8 (31) | 11 (29) | 31 (89)
Tricuspid valve incompetence (Cardiac disorders) | 6 (6) | 1 (1) | 11 (12) | 7 (8) | 25 (27)
Ear discomfort (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (6) | 5 (10)
Ear pain (Ear and labyrinth disorders) | 10 (16) | 7 (8) | 19 (42) | 19 (26) | 55 (92)
Hypoacusis (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 3 (3) | 3 (4) | 8 (10)
Middle ear effusion (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (6)
Vertigo (Ear and labyrinth disorders) | 1 (4) | 2 (2) | 3 (7) | 3 (4) | 9 (17)
Astigmatism (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Conjunctivitis (Eye disorders) | 2 (2) | 2 (2) | 6 (9) | 8 (9) | 18 (22)
Corneal opacity (Eye disorders) | 3 (3) | 5 (5) | 5 (5) | 12 (13) | 25 (26)
Glaucoma (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Myopia (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 3 (4) | 2 (3) | 7 (9)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (5)
Abdominal discomfort (Gastrointestinal disorders) | 3 (6) | 1 (1) | 5 (8) | 7 (18) | 16 (33)
Abdominal distension (Gastrointestinal disorders) | 3 (19) | 0 (0) | 0 (0) | 2 (5) | 5 (24)
Abdominal pain (Gastrointestinal disorders) | 12 (19) | 6 (8) | 22 (59) | 24 (60) | 64 (146)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 8 (15) | 9 (11) | 9 (16) | 18 (72) | 44 (114)
Anal pruritus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Breath odour (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (4) | 7 (7) | 8 (9) | 23 (25)
Dental caries (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 3 (4) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 11 (26) | 11 (27) | 25 (71) | 23 (43) | 70 (167)
Dyspepsia (Gastrointestinal disorders) | 3 (26) | 5 (5) | 3 (5) | 2 (2) | 13 (38)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (6) | 1 (1) | 2 (2) | 1 (1) | 6 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 7 (9)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 5 (7)
Nausea (Gastrointestinal disorders) | 15 (34) | 10 (18) | 26 (65) | 28 (91) | 79 (208)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5)
Toothache (Gastrointestinal disorders) | 3 (4) | 3 (5) | 8 (14) | 4 (4) | 18 (27)
Vomiting (Gastrointestinal disorders) | 20 (105) | 17 (62) | 39 (134) | 38 (160) | 114 (461)
Asthenia (General disorders) | 1 (1) | 2 (2) | 1 (2) | 4 (5) | 8 (10)
Catheter site pain (General disorders) | 2 (6) | 0 (0) | 6 (6) | 5 (12) | 13 (24)
Chest discomfort (General disorders) | 3 (4) | 2 (3) | 2 (2) | 3 (3) | 10 (12)
Chest pain (General disorders) | 1 (1) | 2 (2) | 3 (5) | 4 (4) | 10 (12)
Chills (General disorders) | 4 (4) | 1 (1) | 8 (10) | 9 (14) | 22 (29)
Device dislocation (General disorders) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 6 (7)
Device occlusion (General disorders) | 1 (1) | 1 (3) | 2 (2) | 4 (6) | 8 (12)
Effusion (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 4 (5)
Extravasation (General disorders) | 0 (0) | 3 (3) | 3 (6) | 5 (5) | 11 (14)
Fatigue (General disorders) | 10 (17) | 13 (45) | 16 (32) | 19 (50) | 58 (144)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (3) | 7 (8)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 3 (4) | 5 (5) | 9 (10)
Hyperthermia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 8 (9)
Infusion site extravasation (General disorders) | 3 (4) | 1 (2) | 9 (12) | 4 (4) | 17 (22)
Infusion site pain (General disorders) | 2 (2) | 1 (1) | 6 (8) | 4 (6) | 13 (17)
Infusion site rash (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Infusion site swelling (General disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 6 (6)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (5)
Local swelling (General disorders) | 3 (7) | 0 (0) | 5 (5) | 4 (9) | 12 (21)
Malaise (General disorders) | 2 (2) | 3 (5) | 6 (7) | 3 (5) | 14 (19)
Medical device complication (General disorders) | 2 (2) | 1 (3) | 5 (6) | 5 (8) | 13 (19)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 8 (8)
Oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (4) | 0 (0) | 4 (4) | 3 (4) | 8 (12)
Pain (General disorders) | 5 (6) | 1 (3) | 6 (8) | 5 (7) | 17 (24)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 6 (6)
Pyrexia (General disorders) | 22 (91) | 19 (62) | 38 (113) | 39 (231) | 118 (497)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 5 (8) | 3 (3) | 9 (12)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (4) | 4 (6) | 2 (3) | 10 (15)
Bronchitis (Infections and infestations) | 5 (7) | 3 (4) | 7 (8) | 6 (8) | 21 (27)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 7 (9) | 3 (3) | 5 (13) | 16 (42) | 31 (67)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 7 (7)
Furuncle (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 1 (3) | 3 (7)
Gastroenteritis (Infections and infestations) | 5 (9) | 9 (13) | 24 (36) | 17 (20) | 55 (78)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 7 (7)
Gingivitis (Infections and infestations) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 7 (8)
Hordeolum (Infections and infestations) | 1 (2) | 1 (1) | 6 (14) | 0 (0) | 8 (17)
Influenza (Infections and infestations) | 3 (7) | 5 (6) | 11 (24) | 5 (6) | 24 (43)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (4)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 5 (6) | 6 (8)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 2 (2) | 3 (3) | 7 (8)
Nasopharyngitis (Infections and infestations) | 13 (34) | 13 (28) | 29 (62) | 28 (67) | 83 (191)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 4 (7) | 1 (1) | 6 (9)
Oral herpes (Infections and infestations) | 1 (2) | 1 (1) | 4 (7) | 0 (0) | 6 (10)
Otitis externa (Infections and infestations) | 3 (4) | 1 (1) | 8 (15) | 6 (8) | 18 (28)
Otitis media (Infections and infestations) | 8 (10) | 5 (5) | 11 (29) | 10 (18) | 34 (62)
Otitis media acute (Infections and infestations) | 1 (2) | 2 (2) | 5 (11) | 4 (6) | 12 (21)
Pharyngitis (Infections and infestations) | 9 (12) | 6 (7) | 8 (10) | 11 (18) | 34 (47)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2) | 3 (6) | 3 (4) | 9 (13)
Rhinitis (Infections and infestations) | 9 (21) | 6 (17) | 11 (30) | 9 (19) | 35 (87)
Sinusitis (Infections and infestations) | 5 (7) | 1 (1) | 4 (4) | 4 (6) | 14 (18)
Tinea pedis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Tonsillitis (Infections and infestations) | 2 (3) | 2 (2) | 5 (8) | 6 (7) | 15 (20)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 13 (53) | 8 (25) | 24 (82) | 24 (81) | 69 (241)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 6 (6)
Viral infection (Infections and infestations) | 1 (3) | 3 (5) | 9 (12) | 5 (6) | 18 (26)
Viral pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 6 (12) | 0 (0) | 5 (9) | 5 (10) | 16 (31)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 6 (7) | 9 (10)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (3) | 2 (3) | 7 (9)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 6 (7)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 3 (4) | 12 (20) | 5 (7) | 24 (36)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (8) | 2 (2) | 7 (11)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (5) | 0 (0) | 2 (4) | 2 (3) | 7 (12)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 4 (5)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 6 (6)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 6 (6)
Procedural pain (Injury, poisoning and procedural complications) | 3 (9) | 2 (2) | 6 (7) | 7 (9) | 18 (27)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Blood pressure diastolic increased (Investigations) | 0 (0) | 2 (4) | 3 (9) | 3 (4) | 8 (17)
Blood pressure increased (Investigations) | 2 (6) | 0 (0) | 3 (3) | 1 (1) | 6 (10)
Blood pressure systolic increased (Investigations) | 0 (0) | 2 (7) | 3 (28) | 1 (2) | 6 (37)
Blood urine present (Investigations) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Heart rate decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Heart rate increased (Investigations) | 2 (3) | 1 (1) | 4 (4) | 7 (13) | 14 (21)
Oxygen saturation decreased (Investigations) | 6 (17) | 3 (15) | 9 (16) | 10 (26) | 28 (74)
Respiratory rate increased (Investigations) | 4 (5) | 1 (1) | 2 (2) | 3 (3) | 10 (11)
Vital capacity decreased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 5 (5) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (90) | 16 (57) | 40 (93) | 29 (94) | 105 (334)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (17) | 4 (6) | 19 (45) | 18 (46) | 51 (114)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Knee deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 1 (1) | 6 (6) | 14 (15)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 1 (1) | 3 (4) | 9 (11)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (2) | 5 (5) | 2 (2) | 9 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (14) | 4 (9) | 10 (14) | 9 (20) | 30 (57)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 3 (4) | 1 (1) | 7 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 1 (1) | 3 (3) | 5 (9) | 16 (24)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3) | 9 (14) | 10 (24) | 31 (50)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (54) | 12 (25) | 27 (80) | 31 (102) | 86 (261)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (6) | 8 (9)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Cervical cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 5 (6) | 6 (6) | 8 (20) | 12 (30) | 31 (62)
Headache (Nervous system disorders) | 23 (102) | 16 (67) | 39 (232) | 36 (271) | 114 (672)
Hyperreflexia (Nervous system disorders) | 2 (3) | 3 (4) | 1 (2) | 0 (0) | 6 (9)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 7 (8)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (4) | 8 (9)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 7 (18) | 11 (22)
Somnolence (Nervous system disorders) | 2 (28) | 3 (3) | 1 (1) | 4 (4) | 10 (36)
Syncope (Nervous system disorders) | 0 (0) | 2 (9) | 0 (0) | 1 (1) | 3 (10)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (6) | 7 (9)
Anxiety (Psychiatric disorders) | 3 (4) | 3 (4) | 5 (7) | 1 (1) | 12 (16)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 5 (6)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 7 (7)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 5 (6)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 7 (7)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 3 (4) | 3 (4) | 8 (10)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (11) | 1 (4) | 5 (24) | 3 (9) | 12 (48)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 5 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 5 (12) | 3 (11) | 12 (28)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (62) | 14 (49) | 37 (85) | 28 (70) | 100 (266)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (7) | 12 (33) | 11 (23) | 34 (71)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 4 (8) | 5 (6) | 8 (19) | 20 (42)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (21) | 4 (6) | 15 (24) | 16 (38) | 45 (89)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 3 (3) | 6 (7) | 3 (3) | 15 (23)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 5 (6)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (24) | 11 (16) | 23 (48) | 27 (63) | 74 (151)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 6 (6)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 4 (6)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 4 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7) | 9 (14) | 2 (2) | 19 (26)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (10) | 7 (16) | 14 (24) | 31 (56)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 6 (7)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 9 (9)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (6) | 2 (4) | 9 (14)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (5) | 8 (9)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 2 (3) | 1 (1) | 7 (9)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 5 (6) | 6 (8) | 4 (6) | 20 (30)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (4) | 10 (11)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (6) | 2 (4) | 5 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 5 (6)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 6 (7)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (7) | 8 (10) | 1 (2) | 15 (21)
Erythema (Skin and subcutaneous tissue disorders) | 6 (12) | 3 (4) | 7 (7) | 10 (29) | 26 (52)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 1 (1) | 3 (3) | 9 (11)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (18) | 3 (6) | 8 (28) | 19 (32) | 37 (84)
Rash (Skin and subcutaneous tissue disorders) | 8 (13) | 8 (30) | 15 (61) | 19 (103) | 50 (207)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (3) | 1 (1) | 4 (7)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (1) | 1 (1) | 3 (3) | 6 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (59) | 2 (28) | 5 (87)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 3 (7)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 9 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (38) | 1 (37) | 11 (53) | 12 (33) | 30 (161)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 6 (6)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 2 (2) | 4 (6) | 0 (0) | 7 (9)
Flushing (Vascular disorders) | 1 (3) | 2 (2) | 2 (2) | 5 (8) | 10 (15)
Hot flush (Vascular disorders) | 0 (0) | 2 (6) | 3 (5) | 2 (2) | 7 (13)
Hypertension (Vascular disorders) | 1 (1) | 4 (13) | 6 (28) | 6 (16) | 17 (58)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 3 (6) | 6 (7) | 12 (16)
Pallor (Vascular disorders) | 2 (3) | 2 (2) | 2 (4) | 7 (21) | 13 (30)
Poor venous access (Vascular disorders) | 6 (21) | 5 (10) | 6 (7) | 8 (16) | 25 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes